CLINICAL TRIAL: NCT00195598
Title: Pilot Study of Venlafaxine Extended Release (XR) in the Treatment of Panic Disorder (PD) in Comparison to Paroxetine.
Brief Title: Study Comparing Venlafaxine vs. Paroxetine in Panic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0600B-101359
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Panic Disorders
Keywords: Panic Disorders
MeSH Terms: conditions — Panic Disorder | interventions — Venlafaxine Hydrochloride; Paroxetine

INTERVENTIONS:
Drug: VENLAFAXINE
Drug: Paroxetine

SUMMARY:
The purpose of this pilot study is to evaluate the improvement in social function following therapy with venlafaxine extended release (XR) in the treatment of panic disorder (PD) in comparison to paroxetine. An additional purpose of this pilot study is to obtain the tolerability of using venlafaxine extended release (XR) in the treatment of panic disorder (PD) in comparison to paroxetine.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM IV criteria for Panic Disorder (with or without agoraphobia) for at least 3 months before study day 1.
* Have a minimum of 8 full-symptom panic attacks during the 4 weeks before the screening visit.
* Provide a written informed consent

Exclusion Criteria:

* Treatment with Venlafaxine within 6 months of study day 1, as well Paroxetine
* Known hypersensitivity to Venlafaxine or related compounds as well to Paroxetine.
* Psychopharmacologic drugs within 14 days of study day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the improvement of social function following therapy with Venlafaxine extended release (XR)in the Treatment of Panic Disorder in comparison to Paroxetine.

SECONDARY OUTCOMES:
Obtain the tolerability of using Venlafaxine extended release (XR) in the treatment of Panic Disorder in comparison to Paroxetine.

CONTACTS AND LOCATIONS:
Overall Officials: Trial Manager, Study Director — Pfizer CT.gov Call Center
Locations (3):
- Brazil (3):
  - Jundiaí, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo